CLINICAL TRIAL: NCT07051785
Title: Fruquintinib vs Bevacizumab Combined With Irinotecan Liposome and Capecitabine as Second-Line Therapy for Advanced Metastatic Colorectal Cancer：A Multicenter Randomized Controlled Trial
Brief Title: Fruquintinib vs Bevacizumab Combined With Irinotecan Liposome and Capecitabine as Second-Line Therapy for Advanced Metastatic Colorectal Cancer
Acronym: ARK
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Liu Huang (Other)
Responsible Party: Sponsor-Investigator, Liu Huang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C135
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer (CRC)
Keywords: Colorectal Cancer; Fruquintinib; Second-Line
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fruquintinib+Irinotecan Liposome+Capecitabine (Experimental): fruquintinib(4mg/d, PO, D1-14, Q3W) + irinotecan liposome(56mg/m2, ivgtt, D1, Q3W) + capecitabine(800mg/m2, PO, BID, D1-14, Q3W), every three weeks is a cycle.
  Interventions: Drug: Fruquintinib+Irinotecan Liposome+Capecitabine
- Bevacizumab+Irinotecan Liposome+Capecitabine (Active Comparator): bevacizumab(7.5mg/kg, ivgtt, D1, Q3W)+irinotecan liposome(56mg/m2, ivgtt, D1, Q3W) + capecitabine(800mg/m2, PO, BID, D1-14, Q3W), every three weeks is a cycle.
  Interventions: Drug: Bevacizumab+Irinotecan Liposome+Capecitabine

INTERVENTIONS:
Drug: Fruquintinib+Irinotecan Liposome+Capecitabine — Stage 1: Participants received fruquintinib, irinotecan liposome, and capecitabine for 6-8 cycles. If no disease progression was observed after the initial treatment, patients were transitioned to maintenance therapy with fruquintinib and capecitabine.
  Stage 2: if the primary endpoint of progression-free survival (PFS) was met in the first stage, participants were eligible for the second stage. Participants were randomly assigned to two groups (A and B), Group A: Fruquintinib + irinotecan liposome + capecitabine. After 6-8 cycles of treatment, patients who had no disease progression were transitioned to maintenance therapy with Fruquintinib + capecitabine
  Arms: Fruquintinib+Irinotecan Liposome+Capecitabine
Drug: Bevacizumab+Irinotecan Liposome+Capecitabine — Stage 2: if the primary endpoint of progression-free survival (PFS) was met in the first stage, participants were eligible for the second stage. Participants were randomly assigned to two groups (A and B), Group B: Bevacizumab + irinotecan liposome + capecitabine. After 6-8 cycles of treatment, patients who had no disease progression were transitioned to maintenance therapy with bevacizumab + capecitabine
  Arms: Bevacizumab+Irinotecan Liposome+Capecitabine

SUMMARY:
This study is divided into two phases. The first phase aims to preliminarily evaluate the efficacy and safety of fruquintinib in combination with irinotecan liposome and capecitabine as second-line therapy for advanced metastatic colorectal cancer. The second phase is designed to further assess the efficacy and safety of fruquintinib in combination with irinotecan liposome and capecitabine compared to bevacizumab in combination with chemotherapy, also as second-line treatment for advanced metastatic colorectal cancer.

The first phase is a single-arm study, while the second phase is a randomized (1:1) controlled trial. Entry into the second phase is determined by the investigators based on the efficacy results from the first phase study: if the primary endpoint of progression-free survival (PFS) is met in the first phase, participants will proceed to the second phase study. In the second phase, randomization is stratified according to the RAS status and the presence of disease progression within six months of adjuvant or neoadjuvant therapy.

In the second phase, patients will be ramdomly assigned to receive fruquintinib(4mg/d, PO, D1-14, Q3W) in combination with irinotecan liposome(56mg/m2, ivgtt, D1, Q3W) and capecitabine(800mg/m2, PO, BID, D1-14, Q3W) or bevacizumab(7.5mg/kg, ivgtt, D1, Q3W) in combination with the same chemotherapy. Every three weeks is a cycle.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the most common malignant tumors in the gastrointestinal tract, ranking third globally in terms of incidence and second in terms of mortality. The incidence rate is higher in developed countries compared to developing countries. According to statistical data from the Chinese Cancer Center in 2018, CRC ranks third and fifth in terms of incidence and mortality, respectively. Due to its insidious onset and non-specific clinical manifestations, the early detection rate of CRC is relatively low. Approximately 50% to 60% of patients diagnosed at an advanced stage, often with metastasis.

The treatment of colorectal cancer (CRC) encompasses surgery, chemotherapy, radiotherapy, targeted therapy, and immunotherapy. For patients with early-stage CRC, curative surgery is the primary therapeutic approach; however, recurrence and metastasis remain potential risks. In contrast, for patients with metastatic, unresectable CRC (mCRC), the treatment aims to prolong survival and improve quality of life . According to the guidelines, systemic therapy primarily involves chemotherapy and, in some cases, the combination of chemotherapy and targeted agents . Traditional chemotherapeutic agents include 5-FU, capecitabine, irinotecan, oxaliplatin, and etc.. Commonly used targeted therapies include monoclonal antibodies, such as bevacizumab and cetuximab. The use of these biologics which are blocking key pathways in the progression of mCRC has further prolonged patient survival. However, most patients with unresectable metastatic CRC experience disease progression or develop unacceptable toxicity during first-line systemic therapy, necessitating the initiation of second-line treatment.

The goal of this clinical trial is to evaluate the efficacy and safety of fruquintinib combined with irinotecan liposome and capecitabine as second-line therapy for advanced metastatic colorectal cancer in patients histopathologically confirmed unresectable colorectal cancer, who have previously failed or were intolerant to standard treatment.

This study is a multicenter, two-stage, randomized controlled trial. Participants were enrolled from patients who had previously received standard first-line therapy based on oxaliplatin, which failed or was not tolerated. The study aims to further evaluate the efficacy and safety of the combination of fruquintinib, irinotecan liposome, and capecitabine compared to bevacizumab combined with chemotherapy as second-line treatment for metastatic, unresectable colorectal cancer (mCRC).

Study Design:

Stage 1: Single-Arm Cohort

* A total of 28 patients were enrolled in this phase.
* Participants received fruquintinib, irinotecan liposome, and capecitabine for 6-8 cycles.
* If no disease progression was observed after the initial treatment, patients were transitioned to maintenance therapy with fruquintinib and capecitabine.
* Imaging assessments were conducted every 6 weeks (±7 days), and responses were evaluated according to RECIST 1.1 criteria.

Stage 2: Randomized (1:1) Controlled Trial

* Based on the results of the first stage, investigators determined whether to proceed to the second stage. If the primary endpoint of progression-free survival (PFS) was met in the first stage, participants were eligible for the second stage.
* A total of 40 patients were planned to be enrolled in this phase.
* Randomization was stratified based on RAS mutation status and disease progression within 6 months of adjuvant or neoadjuvant therapy.
* Participants were randomly assigned to two groups (A and B), each consisting of 20 patients:

  * Group A: Fruquintinib + irinotecan liposome + capecitabine
  * Group B: Bevacizumab + irinotecan liposome + capecitabine
* After 6-8 cycles of treatment, patients who had no disease progression were transitioned to maintenance therapy:

  * Group A: Fruquintinib + capecitabine
  * Group B: Bevacizumab + capecitabine
* Imaging assessments were conducted every 6 weeks (±7 days), and responses were evaluated according to RECIST 1.1 criteria

ELIGIBILITY:
Inclusion criteria:

1. Patients voluntarily enrolled in the study and signed an informed consent form, were compliant and cooperated with follow-up visits;
2. Patients with metastatic colorectal adenocarcinoma confirmed by pathology or histology;
3. Age: 18-75 (inclusive of 18 and 75), male or female;
4. Patients who have previously failed or were intolerant to first-line standard therapy (recurrence within 6 months of the end of adjuvant chemotherapy is considered first-line treatment failure).
5. ECOG score: 0-1;
6. At least one measurable lesion (based on RECIST 1.1 criteria);
7. Major organs and bone marrow function were essentially normal (no blood components or cell growth factors had been used in the 14 days prior to enrollment):

   * Neutrophil count ≥ 1.5 × 10⁹/L;
   * Platelet count ≥ 100 × 10⁹/L;
   * Hemoglobin ≥ 90 g/L;
   * Coagulation parameters: International Normalized Ratio (INR) ≤ 1.5 × ULN; Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN;
   * Liver function: Total bilirubin ≤ 1.5 × ULN; Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 2.5 × ULN (with an exception for patients with liver metastases, where ALT/AST may be up to 5 × ULN);
   * Renal function: Serum creatinine ≤ 1.5 × ULN; Creatinine clearance (CCr) ≥ 50 mL/min.
8. Female participants of reproductive age must undergo a serum or urinalysis that shows no pregnancy within 14 days before the first dose of study treatment. Male or female patients of childbearing potential will voluntarily use an effective method of contraception, e.g., double-barrier contraception, condoms, oral or injectable contraceptives, intrauterine devices, etc., during the study period and for at least 6 months after the last dose of study medication.

Exclusion criteria:

1. History of major surgery or severe trauma within 4 weeks prior to the initiation of the study drug.
2. Use of immunosuppressive agents, including systemic or locally absorbed corticosteroids, for immunosuppressive purposes, with a daily dose of prednisone >10 mg or equivalent, and continued us within 2 weeks prior to enrollment.
3. Prior exposure to any irinotecan-containing chemotherapy regimen.
4. Reception of live attenuated vaccines within 4 weeks prior to the initiation of the study drug.
5. Prior treatment with anti-angiogenic small-molecule targeted therapy.
6. Presence of any active autoimmune disease or a history of autoimmune disorders (e.g., autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypopituitarism, vasculitis, nephritis and etc.; not include vitiligo or childhood asthma that has fully resolved and does not require intervention in adulthood; asthma requiring bronchodilator therapy for medical management is included).
7. History of other malignancies within the past 5 years, except for curatively resected skin basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma in situ.
8. Congenital or acquired immunodeficiency (e.g., HIV) or active hepatitis (e.g., hepatitis B: HBsAg positive and HBV DNA ≥ 10⁴ copies/mL or >2000 IU/mL; hepatitis C: HCV antibody positive).
9. Uncontrolled cardiac clinical symptoms or diseases, including: (1) NYHA classification >2 heart failure; (2) Unstable angina pectoris; (3) Myocardial infarction within 1 year; (4) Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.
10. Hypertension that is not well-controlled with antihypertensive medication (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg).
11. Active or uncontrolled severe infections (≥ CTCAE grade 2 infection).
12. Urine routine suggests urinary protein ≥2+ and the amount of urinary protein >1.0g in 24 hours.
13. Patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding >30 mL within 3 months, vomiting blood, black stool, blood in stool), hemoptysis (>5 mL of fresh blood within 4 weeks), or a thromboembolic event (including stroke events and/or transient ischemic attack) within 12 months;
14. Active peptic ulcer disease, ulcerative colitis, or uncontrolled gastrointestinal bleeding, or any gastrointestinal condition judged by the investigator, which may cause gastrointestinal bleeding, perforation, or bowel obstruction.
15. Female participants who are pregnant (positive pregnancy test prior to drug administration) or are breastfeeding;.
16. Patients who are allergic to the study drug or excipients.
17. Any other conditions judged by the investigator which can potentially affect the study outcomes or compromise the safety or adherence of the participants, such as drug abuse, serious diseases (including psychiatric conditions like epilepsy), or other medical, psychological, or social factors that may endanger participant safety or adherence.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-07-07 (Estimated); Primary Completion 2027-07-06 (Estimated); Study Completion 2028-07-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | one year
  time from randomization to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | one year
  the proportion of patients with complete response or partial response, using RECIST v 1.1.
Disease Control Rate (DCR) | one year
  the proportion of patients with complete response, partial response or stable disease, using RECIST v 1.1.
Overall survival (OS) | two years
  time from randomization to death from any cause